CLINICAL TRIAL: NCT00638768
Title: Effectiveness of Physiotherapy for Vertebral Osteoporotic Fracture: a Randomised Controlled Pilot Trial
Brief Title: Effectiveness of Physiotherapy for Osteoporotic Spinal Fracture
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: ANZ Trustees (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 010085.1
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2025-07-10 (Actual); Status verified 2008-03

CONDITIONS: Osteoporosis; Vertebral Fracture
Keywords: physical therapy; rehabilitation; pain; osteoporosis; vertebral fracture
MeSH Terms: conditions — Osteoporosis; Spinal Fractures; Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physiotherapy (Active Comparator): Including 10 individual visits with a physiotherapist and home exercises
  Interventions: Other: Physiotherapy
- 2 (No Intervention): Usual care

INTERVENTIONS:
Other: Physiotherapy — 10 weekly individual sessions with the therapist each lasting approximately 45 minutes. Techniques included postural taping, massage, mobilisation, exercises. The patients also performed home exercises
  Arms: Physiotherapy

SUMMARY:
The aim of this pilot study was to determine the effect of physiotherapy on impairments and health-related quality of life in people with a painful osteoporotic spinal fracture. It is hypothesised that physiotherapy will reduce impairments and improve quality of life in this patient group.

ELIGIBILITY:
Inclusion Criteria:

* if female, at least five years post-menopause
* aged > 50 years
* primary osteoporosis defined as DXA T score < -2.5 at either the spine or proximal femur with at least one morphometric vertebral crush fracture sustained between 3 months to 2 years previously
* back pain/discomfort in thoracic or lumbar region felt at least weekly within the last 6 months
* stable dose of medication for treatment of osteoporosis (eg. hormone replacement therapy, bisphosphonates)
* community dwelling and able to attend for treatment
* English speaking

Exclusion Criteria:

* secondary causes of bone loss such as osteomalacia, glucocorticoid medication etc.
* co-morbidities that would interfere with participation in exercise such as severe heart or pulmonary disease, inflammatory joint disease, severe osteoarthritis, psychiatric condition
* acute vertebral fracture in past 3 months
* signs and symptoms arising from nerve root compression
* back pain radiating into the lower limb
* previous participation in a formal pain management program for back pain
* physiotherapy for back pain in the past 6 months
* allergic reaction to adhesive tape or poor skin condition that would prevent use of tape

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-02-01 (Actual); Primary Completion 2010-01-01 (Actual); Study Completion 2010-02-10 (Actual)

PRIMARY OUTCOMES:
Back pain as assessed by a numeric rating scale | Baseline and 10 weeks

SECONDARY OUTCOMES:
activity restriction, health-related quality of life and physical activity levels as well as overall perceived rating of change in back pain. Objective measures of thoracic kyphosis, standing balance, back and shoulder muscle endurance | Baseline and 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kim L Bennell, PhD, Principal Investigator — University of Melbourne
Locations (1):
- School of Physiotherapy, University of Melbourne, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Bennell KL, Matthews B, Greig A, Briggs A, Kelly A, Sherburn M, Larsen J, Wark J. Effects of an exercise and manual therapy program on physical impairments, function and quality-of-life in people with osteoporotic vertebral fracture: a randomised, single-blind controlled pilot trial. BMC Musculoskelet Disord. 2010 Feb 17;11:36. doi: 10.1186/1471-2474-11-36. PMID 20163739